CLINICAL TRIAL: NCT01143558
Title: Searching for Persistence of Infection in Lyme Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 100139; 10-I-0139
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-03-10

CONDITIONS: Lyme Disease
Keywords: Borrelia Burgdorferi; Xenodiagnosis; Ticks; Skin Biopsy; Lyme Disease
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- 1 (Experimental): All cohorts undergo the same intervention with the study device.
  Interventions: Device: Lyme Disease Xenodiagnosis

INTERVENTIONS:
Device: Lyme Disease Xenodiagnosis — Clean laboratory-bred ticks are the FDA registered IDE. These ticks are placed on patients to search for evidence of Borrelia burgdorferi.

SUMMARY:
Background:

Lyme disease is an infection caused by Borrelia burgdorferi, a bacteria that is transmitted to humans by ticks. It can cause many different symptoms including rash, fever, headache, meningitis (infection of the central nervous system), and arthritis. While most patients improve after taking antibiotics, some patients continue to have symptoms. It is currently unknown why some patients continue to have symptoms. One possibility is that the antibiotics have not successfully gotten rid of all of the bacteria. Current tests for Lyme disease cannot tell whether the bacteria have been successfully eliminated from the body.

Xenodiagnosis is a way to look for Borrelia bacteria using the animal that usually hosts them, Ixodes scapularis (also known as the deer tick). This method takes advantage of the evolution of the bacteria and the insect that transmits the infection, which can make the insect particularly good at finding the agent. In studies of animals, xenodiagnosis may be more sensitive than current tests for detecting the presence of the Lyme disease bacteria. Researchers are interested in using xenodiagnosis to determine whether uninfected ticks that feed on humans who have been infected with Lyme disease bacteria can detect the continued presence of live bacteria.

Objectives:

- To determine whether xenodiagnosis can be used to successfully investigate the presence of Lyme disease bacteria.

Eligibility:

1. Individuals at least 18 years of age who are in one of the following categories:
2. Have had the erythema migrans rash (a symptom of Lyme infection) and received antibiotic therapy less than 4 months ago (but have not had antibiotics in the previous month).
3. Have the erythema migrans rash and received less than 2 days of antibiotic therapy.
4. Have been diagnosed with early or late Lyme disease, have received antibiotic therapy, but still have high levels of antibodies against the bacteria at least 6 months after therapy, and have not received antibiotics in the past 3 months.
5. Have been diagnosed with early or late Lyme disease, have received antibiotic therapy, and have new complaints of fatigue or other symptoms that are persistent for at least 6 months after completion of antibiotic therapy, and have not received antibiotics in the past 3 months.
6. Have been diagnosed with Lyme arthritis and have not yet received antibiotic therapy.
7. Healthy volunteers who have not had Lyme disease will also be included in this study.

Design:

* Participants will have an initial visit for a physical examination, medical history, and blood sample.
* For the first study visit, researchers will place a strip of filter paper or a small plastic container with 20 to 30 disease-free ticks on the participant s skin. If possible, the ticks will be placed at the site of a Lyme disease rash or another suspicious area, or on the nondominant forearm. Participants will be asked to keep the ticks in place, and will keep a diary card at home to record any symptoms or problems.
* The ticks will be collected 4 to 6 days after placement. At that visit, participants will have a skin biopsy taken of the area tested, a blood sample will be collected, and participants will receive a new diary card to keep until the next clinic visit.
* After 1 month, participants will provide a final blood sample, and will receive a follow-up phone call 2 months afterward.

DETAILED DESCRIPTION:
Lyme disease is the most common vector borne disease in the United States. Although antibiotic therapy is clinically effective in treating the symptoms of Lyme disease for most patients early in the course of disease, a significant number of patients who receive therapy report persistent symptoms. The cause of persistent symptoms after antibiotic therapy for Lyme disease is an area of great controversy. Recent studies have shown that the organism (Borrelia burgdorferi) may persist in animals after antibiotic therapy and can be detected by using the natural tick vector (Ixodes scapularis) to acquire the organism through feeding (xenodiagnosis). Whether this occurs in humans is unknown. Currently available tests for human Lyme disease do not allow determination of persistent infection after antibiotic therapy.

In this proposal, the utility of xenodiagnosis for identifying persistence of B. burgdorferi in treated human Lyme disease will be tested in up to 120 subjects with various stages of Lyme disease with 30 healthy adults to serve as controls. Subjects will be followed for approximately 3 months. In Objective #1, subjects who have the characteristic erythema migrans (EM) rash and have been treated with antibiotics early (within 3 weeks of infection) in the course of Lyme disease will be tested. After completion of antibiotic therapy, 25-30 larval Ixodes ticks will be allowed to feed on the subject and biopsies of the EM site will be performed. Repleted ticks will be collected and tested for the presence of B. burgdorferi. In Objective #2, similar studies will be performed, but enrollment will target subjects with elevated C6 (region 6 of the VlsE surface protein of B. burgdorferi) antibody levels. In Objective #3, patients with persistent symptoms after antibiotic therapy will be evaluated. As an attempt to increase the chances of a positive xenodiagnosis in humans, patients with EM who are in the first 2 days of antibiotic therapy and patients with untreated Lyme arthritis will also be evaluated. Evidence that B. burgdorferi can be recovered by xenodiagnosis after antibiotic therapy in subjects with continued symptoms would change the current paradigm for potential mechanisms of disease and provide researchers and clinicians a tool for identifying patients with persistent infection. In Objective #4 we will assess the safety of the planned xenodiagnostic procedure in humans. All individuals who underwent xenodiagnosis under the study will be assessed for adverse events.

ELIGIBILITY:
* INCLUSION CRITERIA:

Criteria for the diagnosis of Lyme disease can be found at The clinical assessment, treatment, and prevention of Lyme disease, human granulocytic anaplasmosis, and babesiosis: clinical practice guidelines by the Infectious Diseases Society of America (4).

1. Patients With EM (N=35), Post Treatment

   * Age 18 or older
   * EM diagnosed by the study physician or, with a diagnosis of EM that is thought to be highly likely by the study physician.
   * Treatment with at least 1 course of antibiotics that fulfills the Infectious Diseases Society of America guidelines for the recommended therapy for Lyme disease. There must be at least 1 month and up to 4 months between the end of the therapy and the study procedures.
2. High C6 Antibody Titer (N=35)

   * Age 18 or older
   * Diagnosed with confirmed or probable early or late Lyme disease as per Centers for Disease Control and Prevention (CDC) case definition (http://www.cdc.gov/ncphi/disss.nndss/caseded/lyme disease 2008.htm), have received recommended antibiotic therapy and have a high C6 ELISA titer (index above 3) at least 6 months after therapy.
3. Post Lyme disease syndrome (N=20)

   * Age 18 or older
   * Diagnosed with confirmed or probable early or late Lyme disease fulfilling the case definition of Lyme disease by the CDC (http://www.cdc.gov/ncphi/disss.nndss/caseded/lyme disease 2008.htm)
   * Received recommended antibiotic therapy, with resolution or stabilization of the objective manifestation(s) of Lyme disease.
   * New complaints of fatigue, paresthesias or dysesthesias, widespread musculoskeletal pain or cognitive difficulties within 6 months of the diagnosis of Lyme disease
   * Symptoms are persistent or relapsing for at least a 6-month period after completion of antibiotic therapy, causing reduction in previous levels of occupational, educational, social, or personal activities.
   * No antibiotic therapy active against Lyme disease in the previous 3 months.
4. Patients With EM (N=20), On Treatment

   * Age 18 or older
   * EM diagnosed by the study physician and receiving antibiotic therapy for less than 48 hours.
5. Lyme Arthritis (N=10)

   * Age 18 or older
   * Lyme arthritis and have not received therapy.
6. Healthy Volunteers (N=30)

   * Age 18 or older
   * No history of Lyme disease
   * Negative whole-cell Borrelia ELISA or C6 ELISA
   * Living in an endemic area for Lyme disease.

EXCLUSION CRITERIA:

* History of allergy to surgical tape or Nitex nylon mesh
* History of severe reactions to tick bites (granuloma or systemic reactions)
* Inability to maintain the dressing for any reason
* Currently receiving any antibiotic or having received antibiotics in the last month (3 months for patients with post Lyme disease syndrome and high C6 titer) (except patients with EM on treatment)
* Pregnancy or lactation
* Unwillingness to use an effective method of birth control for 3 months after tick placement (women of child-bearing potential only)
* Not able to understand all of the requirements of the study or unable to give informed consent and/or comply with all aspects of the evaluation.
* Investigational therapy during the time of the study and/or in the month prior to signing the informed consent.
* Active severe skin disease, uncontrolled diabetes, cancer other than non-melanoma skin cancers, autoimmune disease requiring immunosuppressive therapy, or history of HIV, chronic viral hepatitis, or syphilis.
* Oral steroids in the previous 2 weeks (nasal steroids and replacement doses of steroids are not exclusions)
* Any other condition that, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with the patient participating in and completing the study.

EXCLUSION FROM SKIN BIOPSY PART OF THE PROTOCOL:

* History of forming large thick scars after skin injuries or surgery
* History of excessive bleeding after cuts or procedures
* Currently taking anticoagulants
* History of allergy to lidocaine
* Biopsies will not be done on face, neck, scalp, or over the tibia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-11-04 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
To assess the safety of the planned xenodiagnostic procedure in humans. All individuals who underwent xenodiagnosis under the study will be assessed for adverse events | full duration of the study
  AE reporting per protocol toxicity table
To perform xenodiagnosis on subjects who have the characteristic EM rash and have been treated with antibiotics early in the course of Lyme disease. | Samples collected during tick removal visit.
  PCR and culture of samples
To perform xenodiagnosis on subjects who have a high C6 ELISA titer after antibiotic therapy. | Samples collected during tick removal visit.
  PCR and culture of samples
To perform xenodiagnosis on subjects with post Lyme disease syndrome. | Samples collected during tick removal visit.
  PCR and culture of samples
To perform xenodiagnosis on subjects with newly diagnosed EM lesions that are within 48 hrs of starting antibiotics. | Samples collected during tick removal visit.
  PCR and culture of samples

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Marques, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Tufts University, Boston, Massachusetts

REFERENCES:
- [Background] Bockenstedt LK, Mao J, Hodzic E, Barthold SW, Fish D. Detection of attenuated, noninfectious spirochetes in Borrelia burgdorferi-infected mice after antibiotic treatment. J Infect Dis. 2002 Nov 15;186(10):1430-7. doi: 10.1086/345284. Epub 2002 Oct 23. PMID 12404158
- [Background] Hodzic E, Feng S, Holden K, Freet KJ, Barthold SW. Persistence of Borrelia burgdorferi following antibiotic treatment in mice. Antimicrob Agents Chemother. 2008 May;52(5):1728-36. doi: 10.1128/AAC.01050-07. Epub 2008 Mar 3. PMID 18316520
- [Derived] Marques A, Telford SR 3rd, Turk SP, Chung E, Williams C, Dardick K, Krause PJ, Brandeburg C, Crowder CD, Carolan HE, Eshoo MW, Shaw PA, Hu LT. Xenodiagnosis to detect Borrelia burgdorferi infection: a first-in-human study. Clin Infect Dis. 2014 Apr;58(7):937-45. doi: 10.1093/cid/cit939. Epub 2014 Feb 11. PMID 24523212
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-I-0139.html